CLINICAL TRIAL: NCT03130621
Title: Screening of Hereditary Upper Gastrointestinal Cancer in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Chief physician, Peking University
Other Study IDs: CGOG1012
Record Dates: First submitted 2017-04-22; First posted 2017-04-26 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Improve the Screening Criteria of Chinese Hereditary Upper Gastrointestinal Tumors

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1. propositus：10ml venous blood for germline mutation detection; tumor biospy tissue for somatic mutation detection(optional)
  2. immediate relatives of propositus with Pathogenic mutation or likely-pathogenic mutation：10ml venous blood for germline mutation detection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adenocarcinoma of upper digestive tract: Early-onset carcinomas ; Family History of Malignancy; Special pathological type; MSI or dMMR; Multiple primary malignant tumors;
  Interventions: Diagnostic Test: Gene detection
- Esophageal squamous cell carcinoma: Family History of Malignancy; Multiple primary malignant tumors; MSI or dMMR;
  Interventions: Diagnostic Test: Gene detection

INTERVENTIONS:
Diagnostic Test: Gene detection — Next-generation sequencing

SUMMARY:
Through exploring the specific genetic mutations in the upper gastrointestinal tract tumors with a family history and specific clinical pathological types，we establish a complete family and follow-up system，in order to improve the screening criteria of Chinese hereditary upper gastrointestinal tumors and carry on primary prevention of disease.

ELIGIBILITY:
Inclusion Criteria:

Patients with gastric cancer, esophageal adenocarcinoma, or duodenal adenocarcinoma meet one of the following criteria:

1. age≤30;
2. age≤35，gastric cancer with special pathological types;
3. age≤50，≥one first-degree relative of a malignant tumor;
4. ≥ two first-degree／second-degree relatives of a malignant tumor，and ≥one first-degree relative;
5. have ≥two types of malignancies，and age ≤50 at the first time of diagnosis;
6. MSI or dMMR of tissue specimen;

Patients with esophageal squamous cell carcinomas meet one of the following criteria:

1. ≥ two first-degree／second-degree relatives of a malignant tumor，and ≥one first-degree relative;
2. have ≥two types of malignancies，and age ≤50 at the first time of diagnosis;
3. MSI or dMMR of tissue specimen;

Exclusion Criteria:

* Patients do not meet one of the inclusion criteria;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Upper Gastrointestinal Cancer
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Pedigree analysis | In the first phase of the project, we plan to detect 40-50 families in one year. And in the second phase，we will increase the number of predigree to 200. We hope to finish the phase before 2022.3
  We plan to analyse the families of patients who met the inclusion criterias through gene detection.

SECONDARY OUTCOMES:
somatic mutation landscape of hereditary upper gastrointestinal cancer | We plan to accomplish sample collection, sequencing and data analysis before 2022.3
  By comparing the landscape of somatic mutation of patients with different pathogenic germiline mutation , we want to explore the pathogenesis and molecule mechanism of hereditary upper digestive tract tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No